CLINICAL TRIAL: NCT04673799
Title: A Randomized, Double-blind and Parallel Group Study to Compare the Pharmacokinetics, Immunogenicity and Safety of MV088 and Prolia® in Healthy Adults.
Brief Title: Comparing of the Pharmacokinetics, Immunogenicity and Safety of MV088 and Prolia® in Healthy Adults.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYJT-MV088-I01; CTR20202419 (Other: National Medical Products Administration)
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: randomized、double-blind、parallel-group、single-dosed、positive control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MV088 (Experimental): MV088 injection (60mg) by subcutaneous injection once on the first day
  Interventions: Drug: MV088 injection
- Prolia® (Active Comparator): Prolia® injection (60mg) by subcutaneous injection once on the first day
  Interventions: Drug: Prolia® injection

INTERVENTIONS:
Drug: MV088 injection — MV088 injection (60mg) by subcutaneous injection once on the first day
  Arms: MV088
Drug: Prolia® injection — Prolia® injection (60mg) by subcutaneous injection once on the first day
  Arms: Prolia®

SUMMARY:
A Randomized, Double-blind and Parallel Group Study to Compare the Pharmacokinetics, Immunogenicity and Safety of MV088 and Prolia® in Healthy Adults.

DETAILED DESCRIPTION:
This is a phase I, double center, randomized, double-blind, single dose and parallel group clinical trial . The primary objective is to assess the pharmacokinetic similarity of MV088 and Prolia® in healthy volunteers. The secondary objectives is to assess the similarity of clinical safety and immunogenicity of MV088 and Prolia® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years or ≤65 years, male(including the boundary value).
2. The body weight is within the range of 50~70kg (including the boundary value) and the body mass index（BMI） is within the range of 19.0~26.0kg/m2 (including the boundary value).
3. Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements.
4. The volunteers are able to communicate well with the researchers, understand and comply with the requirements of the study, and are expected to participate in all follow-up visits (no long-term plans to leave the study site).

Exclusion Criteria:

1. Have participated in any drug or medical device trials or are participating in other clinical trials within 3 months prior to first administration.
2. Occurred or suffering from osteomyelitis or ONJ (mandibular necrosis) previously.
3. The dental or jaw disease that is active, requiring oral surgery; or planned for invasive dental surgery during the study; or dental or oral surgery wounds have not healed.
4. Occurred or suffering hypocalcemia.
5. Have taken any medicine (including Chinese herbal medicine) within 14 days before the first administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-02-22 (Estimated); Primary Completion 2021-10-18 (Estimated); Study Completion 2021-10-18 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of MV088/Prolia in plasma: Cmax | 126 days
  To characterize the pharmacokinetic parameters#Cmax of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: AUC0-∞ | 126 days
  To characterize the pharmacokinetic parameters#AUC0-∞ of MV088/Prolia after the first day administer

SECONDARY OUTCOMES:
Pharmacokinetics of MV088/Prolia in plasma: AUC0-t | 126 days
  To characterize the pharmacokinetic parameters#AUC0-t of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: Tmax | 126 days
  To characterize the pharmacokinetic parameters#Tmax of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: t1/2 | 126 days
  To characterize the pharmacokinetic parameters#t1/2 of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: CLz/F | 126 days
  To characterize the pharmacokinetic parameters#CLz/F of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: Vz/F | 126 days
  To characterize the pharmacokinetic parameters#Vz/F of MV088/Prolia after the first day administer
Pharmacokinetics of MV088/Prolia in plasma: λz | 126 days
  To characterize the pharmacokinetic parameters#λz of MV088/Prolia after the first day administer
Safety evaluation of MV088/Prolia | 126 days
  To characterize the Safety evaluation of MV088/Prolia after the first day administer
Immunogenicity evaluation of MV088/Prolia | 126 days
  To characterize the Immunogenicity evaluation of MV088/Prolia after the first day administer

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, ph.D, Principal Investigator — The Third Hospital of Changsha; Jianchang He, ph.D, Principal Investigator — Yunnan Provincial Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No